CLINICAL TRIAL: NCT02851966
Title: Use of Semen TEX101 to Improve Sperm Retrieval Rates for Men With Non-obstructive Azoospermia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Weill Medical College of Cornell University (Other); McGill University (Other); University of California, San Francisco (Other); The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CAN-TEX-P1
Record Dates: First submitted 2016-07-11; First posted 2016-08-02 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Non-obstructive Azoospermia
Keywords: Non-obstructive Azoospermia; Sperm Retrieval; Infertility, Male; Semen; Biomarkers; Proteomics; Enzyme-Linked Immunosorbent Assay
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TEX101 (Other): This is a single arm study. All patients will be asked to provide multiple semen samples and all samples will be tested with TEX101 ELISA assay. Timing of mTESE maybe changed according to the assay results.
  Interventions: Procedure: mTESE

INTERVENTIONS:
Procedure: mTESE — mTESE time may be postponed or advanced.

SUMMARY:
The investigators hypothesize that sperm production varies with time in men with no sperm in semen (non-obstructive azoospermia, NOA) and that the semen protein, TEX101, is able to monitor these changes. The investigators further hypothesize that TEX101 levels may be used to predict the optimum time for microsurgical testicular sperm extraction (mTESE) to provide the highest successful rates of sperm retrieval.

DETAILED DESCRIPTION:
This is a non-randomized pilot study. All men with NOA, who may or may not consider having mTESE, will be approached to enter this study.

Recruited men will have a semen test performed at the initial visit (time 0) to measure semen TEX101 levels using an ELISA assay.

For men who are not considering a mTESE to retrieve sperm, the TEX101 semen levels will be measured monthly for three months to determine the variability of semen TEX101.

For men who are considering a mTESE in an attempt to retrieve sperm, the mTESE procedure to retrieve sperm will be booked. If the level of TEX101 is detectable at time 0, then the men will have semen testing monthly. If the TEX101 is persistently detectable then the men will have surgery at the time originally scheduled. If the TEX101 drops on any subsequent test to be undetectable, then the semen testing for TEX101 will continue monthly for a maximum of 3 additional months. If the TEX101 remains undetectable for all tests, the men will have the mTESE at the end of the additional 3 months. If the TEX101 is detectable on a subsequent test, then the men will undergo an immediate mTESE (< 2 weeks).

If the initial TEX101 is undetectable, then the men will have monthly semen testing for TEX101 for a maximum of 3 additional tests. If the TEX101 remains persistently undetectable, then a mTESE will be performed as originally booked. If the TEX101 is detected on a subsequent test, then an immediate mTESE (< 2 weeks) is performed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with NOA by standard clinical means with a minimum of 2 semen tests confirming that the man is azoospermic
* Ability to understand the study and consent
* Ability to deliver semen samples

Exclusion Criteria:

* Men do not have NOA
* Cannot understand the study and consent
* Cannot provide semen samples

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-02; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Successful testicular sperm retrieval | 2 years
  This outcome will be measured by if sperms would be found during the procedure or if sperms would be identified in the IVF clinic.

SECONDARY OUTCOMES:
Natural variation in sperm counts in semen | 2 years
  Variation in sperm concentration in semen as measured by direct microscopic assessment of different semen samples provided by each of the participants.
Natural variation in semen TEX101 concentration | 2 years
  Variation in TEX101 concentrations in semen of different semen samples provided by each of the participants as measured by the TEX101 ELISA assay.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Jarvi, MD, Principal Investigator — Mount Sinai Hospital, Canada
Locations (3):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Weill Cornell Medical College, New York, New York
- St. Mary's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided